CLINICAL TRIAL: NCT06140212
Title: Exploring the Relationship Between the Integrated Care for Older People (ICOPE) Framework and Frailty Among Community-dwelling Elderly Individuals
Brief Title: Exploring the Relationship Between ICOPE Framework and Frailty Among Community-dwelling Elderly Individuals
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202310067RINC
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2023-11

CONDITIONS: Community-dwelling Elderly
Keywords: Frailty; ICOPE; Intrinsic capacity; Community-dwelling elderly
MeSH Terms: conditions — Frailty | interventions — Mental Status and Dementia Tests; Self Administration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Decline ICOPE group: The elderly individuals who have at least one impairment in ICOPE screening domains.
  Interventions: Behavioral: Montreal Cognitive Assessment (MoCA); Behavioral: Chinese ICOPE screening tool (self-administration and interview versions); Behavioral: Frailty status assessment (Edmonton frail scale and Frailty criteria by Dr. Fried)
- Non-decline ICOPE group: The elderly individuals who do not have any impairment in ICOPE screening domains.
  Interventions: Behavioral: Montreal Cognitive Assessment (MoCA); Behavioral: Chinese ICOPE screening tool (self-administration and interview versions); Behavioral: Frailty status assessment (Edmonton frail scale and Frailty criteria by Dr. Fried)

INTERVENTIONS:
Behavioral: Montreal Cognitive Assessment (MoCA) — MoCA would be used to assess participants cognitive functioning.
Behavioral: Chinese ICOPE screening tool (self-administration and interview versions) — The ICOPE screening tool would be used to assess participants health status, including cognitive decline, auditory and visual capabilities, mobility restrictions, nutritional status, and depressive symptoms.
Behavioral: Frailty status assessment (Edmonton frail scale and Frailty criteria by Dr. Fried) — The Edmonton frail scale and Frailty criteria by Dr. Fried would be used to assess participants frailty status.

SUMMARY:
This study aims to (1) compare the assessment outcome of the ICOPE-I and ICOPE-S, and (2) investigate the correlation between both versions of the ICOPE step 1 screening tools and frailty in Taiwan.

DETAILED DESCRIPTION:
The prevalence of frailty among the elderly increases annually as the population ages. The World Health Organization (WHO) has introduced the Integrated Care for Older People (ICOPE) framework, which aims to support healthy aging by evaluating the intrinsic capacity (IC) of the elderly in six different areas. In Taiwan, two versions of the ICOPE step 1 screening tools are available: an interview-based version (ICOPE-I) and a self-administered version (ICOPE-S) based on the WHO's model. There are two main models for frailty status assessments: Dr. Fried's phenotype of frailty and Dr. Rockwood's accumulation of deficit models. A comparative study is necessary to assess the consistency of both versions of ICOPE in Taiwan and their associations with frailty.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old
* Community-dwelling elderly
* Walking independently (with/without assistive devices)

Exclusion Criteria:

* Participants with a MoCA score < 26
* Being unable to give informed consent (e.g., aphasia, deafness, and blindness)
* Being unable to finish all the physical and screening assessment assessments

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Communities in Taipei city
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2023-12-02 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Intrinsic capacity | The ICOPE screening tool assessment would take about 10 minutes
  ICOPE screening tool (self-administration and interview version) would be used to evaluate the intrinsic capacity(IC), including cognitive decline, auditory and visual capabilities, mobility restrictions, nutritional status, and depressive symptoms) of the participants.
  Each question requires a binary response, either 'yes' or 'no'. A "total score" will be determined by summing the number of IC impairments, which have a score range of 0-6, with higher scores indicating a greater degree of impairment.
Phenotype of frailty status | The phenotype of frailty status assessment would take about 10 minutes
  Frailty criteria by Dr. Fried would be used to evaluate the frail status of the participants.The Dr. Fried phenotype of frailty comprises five components, unintentional weight loss, exhaustion, weakness, slowness, and low activity. Individuals who exhibit three or more indicators are classified as frail, those with one to two indicators are categorized as pre-frail, and those with no indicators are characterized as robust.
Accumulated frailty status | The accumulated frailty status assessment would take about 10 minutes
  Edmonton frail scale(EFS) would be used to evaluate the frail status of the participants. EFS assesses a wide range of nine domains through 11 questions. These domains cover cognition, general health status, functional independence, social support, medication use, nutrition, mood, continence, and functional performance. The total score of EFS ranges from 0 to 17, where scores of 0-5 indicate not being frail, 6-7 indicate being vulnerable, 8-9 indicate mild frailty, 10-11 indicate moderate frailty and 12-17 indicate severe frailty.

SECONDARY OUTCOMES:
Cognitive status | The cognitive status assessment would take about 10 minutes
  MoCA would be used to evaluate the cognitive functioning of the participants. MOCA comprises attention and concentration, executive function, memory, language ability, visuospatial construction, abstract concepts, calculation, and orientation. The cumulative score amounts to 30 points, with a minimum standard of 26 points or higher. 25-18 points indicate mild cognitive impairment, 17-10 points indicate moderate cognitive impairment, fewer than 10 points indicate severe cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, PhD, Study Chair — National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Zhongzheng, Taiwan